CLINICAL TRIAL: NCT05932940
Title: Incidence of Descemet Membrane Detachment Post Gonioscopy-Assisted Transluminal Trabeculotomy by Anterior Segment Optical Coherence Tomography in Patients With Open Angle Glaucoma
Brief Title: Incidence of Descemet Membrane Detachment Post GATT by AS OCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Elsayed Soliman Ahmed, Opthalmology resident Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-275-2022
Record Dates: First submitted 2023-05-07; First posted 2023-07-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Angle Glaucoma Open
Keywords: gonioscopy-assisted transluminal trabeculotomy; Descemet membrane detachment
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: detection of incidence of Descemet membrane detachment post gonioscopy-assisted transluminal trabeculotomy by anterior segment optical coherence tomography in patients with open angle glaucoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GATT group (Experimental): detection of incidence of Descemet membrane detachment post gonioscopy-assisted transluminal trabeculotomy by anterior segment optical coherence tomography in patients with open angle glaucoma.
  Interventions: Procedure: Gonioscopy-Assisted Transluminal Trabeculotomy

INTERVENTIONS:
Procedure: Gonioscopy-Assisted Transluminal Trabeculotomy — Ab interno angle surgery one of MIGS to lower IOP

SUMMARY:
detection of Incidence of Descemet membrane detachment post gonioscopy-assisted transluminal trabeculotomy by anterior segment optical coherence tomography in patients with open angle glaucoma.

DETAILED DESCRIPTION:
In our study, which should include 30 eyes with OAG who underwent 360 GATT Screening for Descemet Membrane Detachment will be done by Anterior Segment Optical coherence Tomography using SD-OCT: Optovue RTVue (Optovue Inc., Fremont, CA, USA) for the angle day 1 post operative for all patients and 1 week post operative in cases with Descemet membrane detachment to check for spontaneous resolution.

One month post-operative the patients underwent

* Best corrected visual acuity (BCVA) using decimal.
* IOP measurement using GAT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 70 years.
2. Patients with open angle glaucoma undergoing gonioscopy assisted transluminal trabeculotomy.

Exclusion Criteria:

1. Patients with with open angle glaucoma and aphakia.
2. Patients with Congenital Glaucoma.
3. Patients with open angle glaucoma undergoing phaco -gonioscopy-assisted transluminal trabeculotomy.
4. Patients with neovascular glaucoma.
5. Patients with pigmentary Glaucoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Descemet Membrane detachment post GATT | 4 months
  Incidence of Descemet membrane Detachment post Gonioscopy-Assisted Transluminal Trabeculotomy

SECONDARY OUTCOMES:
Amount of reduction of IOP and Glaucoma NGM | 4 months
  Amount of reduction of intraocular pressure and Number of Glaucoma medications
Incidence of Hyphema post GATT | 4 months
  Incidence of Hyphema post Gonioscopy-Assisted Transluminal Trabeculotomy
Incidence of Descemet membrane detachment post gonioscopy-assisted transluminal trabeculotomy by anterior segment optical coherence tomography in patients with open angle glaucoma. | 4 months
  Incidence of Descemet membrane detachment post gonioscopy-assisted transluminal trabeculotomy by anterior segment optical coherence tomography in patients with open angle glaucoma.

CONTACTS AND LOCATIONS:
Overall Officials: Fayrouz Aboalazayem, phD, Principal Investigator — Cairo University
Locations (1):
- Facility of medicine , Cairo University, Cairo, Almanial, Egypt

IPD SHARING:
Plan to Share IPD: No